CLINICAL TRIAL: NCT04299152
Title: Clinical Application of Stem Cell Educator Therapy for the Treatment of Viral Inflammation Caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Brief Title: Stem Cell Educator Therapy Treat the Viral Inflammation in COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Throne Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-TH-001
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Severe Acute Respiratory Syndrome (SARS) Pneumonia
Keywords: severe acute respiratory syndrome coronavirus; Immune modulation; Stem Cell Educator therapy
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia

STUDY DESIGN:
Intervention Model Description: This is a prospective, two-arm, partially masked, single center clinical study to assess the safety, feasibility, and efficacy of SCE therapy for the treatment of patients with SARS-CoV-2.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Stem Cell Educator therapy treat patients with SARS-CoV-2 (Experimental): SCE therapy circulates a patient's blood through a blood cell separator, briefly cocultures the patient's immune cells with adherent CB-SC in vitro, and returns the "educated" autologous immune cells to the patient's circulation.
  Interventions: Combination Product: Stem Cell Educator-Treated Mononuclear Cells Apheresis
- Conventional treatment of patients with SARS-CoV-2 (No Intervention): Patients will receive the regular treatments by only addressing their symptoms such as reducing fever and cough.

INTERVENTIONS:
Combination Product: Stem Cell Educator-Treated Mononuclear Cells Apheresis — SCE therapy circulates a patient's blood through a blood cell separator, briefly cocultures the patient's immune cells with adherent CB-SC in vitro, and returns the "educated" autologous immune cells to the patient's circulation.
  Arms: Stem Cell Educator therapy treat patients with SARS-CoV-2

SUMMARY:
Currently, the growing epidemic of a new coronavirus infectious disease (Covid-19) is wreaking havoc worldwide, which is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). SARS-CoV-2 is a RNA virus that display high similarity in both genomic and proteomic profiling with SARS-CoV that first emerged in humans in 2003 in China. Therefore, preventing and controlling the pandemic occurrences are extremely urgent as a global top priority. Due to the lack of effective antiviral drugs, patients may be treated by only addressing their symptoms such as reducing fever. Clinical autopsies from SARS-CoV-infected patients demonstrated that there were major pathological changes in the lungs, immune organs, and small systemic blood vessels with vasculitis. However, the detection of SARS-CoV were primarily found in the lung and trachea/bronchus, but was undetectable in spleen, lymph nodes, bone marrow, heart and aorta, highlighting the overreaction of immune responses induced by viral infection were really harmful, resulting in the pathogenesis of lungs, immune organs, and small systemic blood vessels. To this respect, immune modulation strategy may be potentially beneficial to enhance anti-viral immunity and efficiently reduce the viral load, improve clinical outcomes, expedite the patient recovery, and decline the rate of mortality in patients after being infected with SARS-CoV-2. Tianhe Stem Cell Biotechnologies Inc. has developed a novel globally-patented Stem Cell Educator (SCE) technology designed to reverse the autoimmune response in Type 1 diabetes (T1D), Alopecia Areata (AA) and other autoimmune diseases. SCE therapy uses human multipotent cord blood stem cells (CB-SC) from human cord blood. Their properties distinguish CB-SC from other known stem cell types, including mesenchymal stem cells (MSC) and hematopoietic stem cells (HSC). Several clinical studies show that SCE therapy functions via CB-SC induction of immune tolerance in autoimmune T cells and restore immune balance and homeostasis in patients with T1D, AA and other inflammation-associated diseases. To correct the overreaction of overreaction of immune responses, the investigators plan to treat SARS-CoV-2 patients with Stem Cell Educator therapy.

DETAILED DESCRIPTION:
This is a prospective, two-arm, partially masked, single center clinical study to assess the safety, feasibility, and efficacy of SCE therapy for the treatment of patients with SARS-CoV-2 infection. Patients will be evaluated by the study principal investigator or co-investigators. Informed consent will be obtained at the initial screening visit. Subjects who meet all criteria will be scheduled for treatment. All enrolled subjects will receive one treatment with the SCE therapy consisting of a single session of mononuclear cells (MNC) collection by apheresis of blood. The MNC product will be treated with the SCE, and followed by an infusion intravenously back to the patient. The SCE-treated subjects will be evaluated according to the schedules of follow-up studies within 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years)
2. Must have a clinical diagnosis of SARS-CoV-2, with at least one of clinical symptoms (e.g., fever ≥38°C, fatigue, cough) and a positive result by the reverse-transcription polymerase chain reaction (RT-PCR) testing
3. Patients must not have received any antiviral treatments known to affect SARS-CoV-2
4. Patients must agree that they are not permitted to use any other treatment to affect SARS-CoV-2 during a period of 6 months after undergoing SCE therapy
5. Adequate venous access for apheresis
6. Ability to provide informed consent
7. For female patients only, willingness to use FDA-recommended birth control (http://www.fda.gov/downloads/ForConsumers/ByAudience/ForWomen/FreePublications/UCM356451.pdf) until 6 months post treatment.
8. Must agree to comply with all study requirements and be willing to complete all study visits

Exclusion Criteria:

1. AST or ALT 2 > x upper limit of normal.
2. Abnormal bilirubin (total bilirubin > 1.2 mg/dL, direct bilirubin > 0.4 mg/dL)
3. Creatinine > 2.0 mg/dl.
4. Known coronary artery disease or EKG suggestive of coronary artery disease unless cardiac clearance for apheresis is obtained from a cardiologist.
5. Known active infection such as Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV)
6. Pregnancy assessed by a positive serum pregnancy test or breastfeeding mothers
7. Use of immunosuppressive medication within one month of enrollment including but not limited to cyclosporine, tacrolimus, sirolimus, and chemotherapy.
8. Anticoagulation other than ASA.
9. Hemoglobin < 10 g/dl or platelets < 100 k/ml
10. Is unable or unwilling to provide informed consent
11. Presence of any other physical or psychological medical condition that, in the opinion of the investigator, would preclude participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-10 (Estimated); Primary Completion 2022-04-09 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Determine the number of Covid-19 patients who were unable to complete SCE Therapy | 4 weeks
  The feasibility will be evaluated by the number of Covid-19 patients who were unable to complete SCE Therapy.

SECONDARY OUTCOMES:
Examine the percentage of activated T cells after SCE therapy by flow cytometry | 4 weeks
  Measurements of immune markers' changes will be preformed by flow cytometry such as activated T cells. Peripheral blood mononuclear cells (PBMC) will be collected at 1, 3, 6, 9, 12, 28 day post the SCE therapy.
Assess the percentage of Th17 cells after SCE therapy by flow cytometry | 4 weeks
  Measurements of immune marker's changes will be preformed by flow cytometry such as the percentage of Th17 cells. Peripheral blood mononuclear cells (PBMC) will be collected at 1, 3, 6, 9, 12, 28 day post the SCE therapy.
Chest imaging changes by computed tomography (CT) scan of the chest | 4 weeks
  Patients will be monitored for their chest imaging every 3 - 5 days for 4 weeks after receiving SCE therapy.
Quantification of the SARS-CoV-2 viral load by real time RT-PCR | 4 weeks
  To determine the viral load by real time RT-PCR, samples of blood, sputum, nose / throat swab will be collected from patients during the follow-up studies after receiving SCE therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Li, MD,PhD, Study Director — Throne Biotechnologies Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Background] Zhao Y. Stem cell educator therapy and induction of immune balance. Curr Diab Rep. 2012 Oct;12(5):517-23. doi: 10.1007/s11892-012-0308-1. PMID 22833322
- [Background] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Zhou H, Yin Z, Chen Y, Zhang Y, Wang S, Shen J, Thaker H, Jain S, Li Y, Diao Y, Chen Y, Sun X, Fisk MB, Li H. Targeting insulin resistance in type 2 diabetes via immune modulation of cord blood-derived multipotent stem cells (CB-SCs) in stem cell educator therapy: phase I/II clinical trial. BMC Med. 2013 Jul 9;11:160. doi: 10.1186/1741-7015-11-160. PMID 23837842
- [Background] Li Y, Yan B, Wang H, Li H, Li Q, Zhao D, Chen Y, Zhang Y, Li W, Zhang J, Wang S, Shen J, Li Y, Guindi E, Zhao Y. Hair regrowth in alopecia areata patients following Stem Cell Educator therapy. BMC Med. 2015 Apr 20;13:87. doi: 10.1186/s12916-015-0331-6. PMID 25896390
- [Background] Delgado E, Perez-Basterrechea M, Suarez-Alvarez B, Zhou H, Revuelta EM, Garcia-Gala JM, Perez S, Alvarez-Viejo M, Menendez E, Lopez-Larrea C, Tang R, Zhu Z, Hu W, Moss T, Guindi E, Otero J, Zhao Y. Modulation of Autoimmune T-Cell Memory by Stem Cell Educator Therapy: Phase 1/2 Clinical Trial. EBioMedicine. 2015 Nov 5;2(12):2024-36. doi: 10.1016/j.ebiom.2015.11.003. eCollection 2015 Dec. PMID 26844283
- [Background] Zhao Y, Jiang Z, Delgado E, Li H, Zhou H, Hu W, Perez-Basterrechea M, Janostakova A, Tan Q, Wang J, Mao M, Yin Z, Zhang Y, Li Y, Li Q, Zhou J, Li Y, Martinez Revuelta E, Maria Garcia-Gala J, Wang H, Perez-Lopez S, Alvarez-Viejo M, Menendez E, Moss T, Guindi E, Otero J. Platelet-Derived Mitochondria Display Embryonic Stem Cell Markers and Improve Pancreatic Islet beta-cell Function in Humans. Stem Cells Transl Med. 2017 Aug;6(8):1684-1697. doi: 10.1002/sctm.17-0078. Epub 2017 Jul 7. PMID 28685960
- See also: Throne Biotechnologies Inc — https://thronebio.com/